CLINICAL TRIAL: NCT06007508
Title: Early Administration of Insulin Glargine in Patients With Diabetic Ketoacidosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study intervention was adopted as standard of care.
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X1935200
Record Dates: First submitted 2022-12-15; First posted 2023-08-23 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-01

CONDITIONS: DKA
Keywords: DKA; Hypoglycemia; Rebound Hyperglycemia; Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: This will be a two arm, prospective, randomized, open label trial in patients presenting with DKA. Block randomization will be used to ensure equal group sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (No Intervention): Subjects presenting to ED with diagnosis of DKA and receiving intravenous short acting insulin will not have orders for subcutaneous insulin glargine placed for research purposes.
- Intervention (Active Comparator): Subjects presenting to ED with diagnosis of DKA will receive study medication set to begin within 2 hours after initiation of the IV insulin infusion. The dose will come from IV pharmacy and dispensed in a 1 mL insulin syringe. If the patient was not taking basal insulin prior to admission, the patient will receive 0.2 units/kg insulin glargine. If the patient was taking basal insulin prior to admission, the patient will receive their home insulin glargine dose.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — Long-acting insulin
  Other Names: Lantus; Basaglar; Semglee
  Arms: Intervention

SUMMARY:
Diabetic ketoacidosis (DKA) is a medical emergency that is associated with significant morbidity and mortality for both patients with type I and type II diabetes. By correcting hyperglycemia and inhibiting the release of free fatty acids, insulin administration leads to decreased ketone formation and resolution of acidosis. Short-acting intravenous insulin is often preferred to subcutaneous administration for initial management due to its short half-life and ease of titration, but patients will eventually need to transition to subcutaneous insulin prior to discharge. The timing of initiation or resumption of home long-acting subcutaneous insulin is controversial in the treatment of DKA. It is currently unknown if resuming a portion or all of the patient's home basal regimen during the initial treatment phase of DKA will provide an impact on patient care. The purpose of this study is to evaluate the impact of early glargine administration if the patient was not previously on basal insulin or resuming the patient's home basal insulin regimen within two hours after the start of the intravenous insulin infusion in addition to usual care will improve patient outcomes.

DETAILED DESCRIPTION:
In 2014, there were 168,000 hospitalizations for DKA, and the average length of stay was 3.4 days in 2009. The estimated annual direct medical expense and indirect cost is 2.4 billion dollars per year. DKA is a potentially life-threatening condition due to its ability to cause metabolic acidosis, electrolyte imbalances, and dehydration. While DKA treatment protocols differ from institution to institution, the goals of treatment remain the same --- resolution of acidosis, dehydration, and hyperglycemia. Following fluid resuscitation, correction of hyperglycemia with insulin therapy is the mainstay of treatment. Intravenous (IV) insulin infusions with regular insulin are commonly used due to its short half-life of 30 to 60 minutes and resulting titratability. Treatment is then continued with subcutaneous (SC) insulin once the acidosis and anion gaps have cleared and the patient's hemodynamics and electrolytes abnormalities have resolved.

Traditionally, when SC insulin is initiated, the IV insulin infusion is stopped two hours later. However, the timing of SC initiation has becoming more controversial in recent years. The 2019 American Diabetes Association Standards of Care recommend transition of patients from IV to SC insulin requires administration of basal insulin 2-4 h prior to the intravenous insulin being stopped to prevent recurrence of ketoacidosis and rebound hyperglycemia. However, the 2014 Joint British Diabetes Societies Inpatient Care Group recommend continuing a patient's home basal insulin during the initial management of DKA to prevent rebound hyperglycemia and to avoid extending length of stay. Several recent papers have examined early basal insulin administration as adjunct therapies with IV insulin infusions for the treatment of hyperglycemia and DKA.

In 2012, a single-center prospective, randomized controlled trial by Hsia et al. compared IV insulin infusion with or without early administration of insulin glargine (dose = 0.25 U/kg) in 61 hyperglycemic patients with diabetes. Forty-one percent (25/61) of the patients enrolled in the trial were admitted with DKA. Those patients that received early glargine had lower prevalence of rebound hyperglycemia when the insulin infusion was discontinued (experimental group: 33% vs control group: 93.5%; P < 0.001). The total length of IV insulin infusion was similar in the two groups (control group: 35 ± 13h vs experimental group: 42 ± 24h). The mean blood glucose levels within the 12-hour study period were significantly lower in the intervention group, while there were 3 asymptomatic hypoglycemic measurements in the control group and none in the intervention group.

In 2015, Doshi et al. conducted a two-center prospective, randomized controlled trial of 40 patients admitted for DKA. Patients were randomized to receive early insulin glargine (dose = 0.3 U/kg) or no glargine in addition to regular care. Those in the early insulin glargine arm were to receive the glargine subcutaneous injection within 2 hours of diagnosis. Patients in the control group were given insulin glargine once the anion gap closed and the IV insulin infusion was continued for two additional hours. There was no difference in time to anion gap closure, hospital length of stay, ICU admissions, ICU length of stay, and hypoglycemic events.

In 2015, Houshyar et al. conducted a single-center, prospective, randomized controlled trial of 40 patients admitted for DKA. Patients were randomized to receive early insulin glargine (dose = 0.4 U/kg) or no insulin glargine in addition to usual care. Patients in the control group were given insulin glargine once the anion gap closed. There was no difference in duration of acidosis, hospital length of stay or rates of hypoglycemia. There were higher rates of hyperglycemia following discontinuation of the insulin infusion in those that did not receive early glargine (51% vs. 35% of measurements in the experimental group showed a glucose >8.3 mM or >150 mg/dL; p = 0.046).

Rappaport et al. (2019) conducted a single-center, retrospective cohort study of 106 admissions for DKA comparing early vs late initiation of basal insulin. Patients admitted to the MICU who were treated with home-dose basal insulin prior to DKA resolution and within 24 hours of IV insulin infusion initiation (n = 33) were compared to patients who were initiated on basal insulin within 6 hours before or any time after IV insulin infusion discontinuation (n = 73). There was no difference in transitional failure, rebound hyperglycemia, hypoglycemia events, time to anion gap closure, length of ICU stay, or hospital length of stay. There was a statistically significant decrease for time on IV insulin infusion (early: 13.8h vs late: 17.1h, p = 0.04).

As previously outlined, randomized studies using weight based basal insulin doses have shown that the early initiation of basal insulin can prevent rebound hyperglycemia with no increase in hypoglycemia. One retrospective study demonstrated a decrease of time on IV insulin infusion in those that received early basal insulin when compared to those that did not. These studies have also shown trends toward shorter ICU and hospital length of stay, anion gap closure, and time to resolution of acidosis but none have demonstrated statistical significance. However, no prospective trials have examined resuming the patient's home basal insulin early in the course of DKA and it is currently unknown if resuming a portion or the entirety of the patient's home basal regimen will provide an impact on patient care.

By conducting a prospective study comparing initiation of early glargine administration at the patient's home dose to current standards of care, early administration may lead to shorter ICU and hospital lengths of stay as well as shorter duration of acidosis. This could provide significant cost-savings to the institution and benefit patients in need of treatment for this serious complication of diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Presented to Regions Hospital ED for chief complaint of DKA, nausea, vomiting, abdominal pain, hyperglycemia, or similar
2. Meets all below diagnostic criteria for DKA per the American Diabetes Association:

   * Arterial or venous pH </= 7.3
   * Serum Bicarbonate </= 18 mEq/L
   * Ketonuria or ketonemia
   * Anion Gap > 10
   * Blood sugar > 250 mg/dL
3. Receiving IV insulin infusion
4. It is feasible to provide insulin glargine within 2 hours (+/- 30 minutes) of IV infusion start
5. Will be admitted to the ICU for DKA, or already admitted to the ICU for DKA
6. Ability to provide informed consent

Exclusion Criteria:

1. Age < 18
2. End stage renal disease or hepatic disease
3. Hypotension requiring IV vasopressors or inotropes at any point during admission (i.e. norepinephrine, dobutamine, vasopressin, etc.)
4. Need for emergent surgery
5. Pregnant patients
6. Prisoners
7. Indication for insulin therapy other than DKA (hypertriglyceridemia, beta-blocker overdose, hyperglycemia without DKA)
8. Patients receiving prior to admission insulin pump therapy
9. Patients receiving prior to admission combination insulin products (i.e. Novolin® 70/30, Novolog® 70/30, Humalog® 75/25, etc.)
10. Did not consent to study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Does early administration of insulin glargine result in a change in ICU length of stay when compared to usual care for the treatment of diabetic ketoacidosis? | Assessed from time of intervention until discharge from ICU to general medical unit or from hospital, up to 12 weeks
  Hypothesis: Early administration of insulin glargine will result in shorter ICU length of stay when compared to usual care in patients with DKA.

SECONDARY OUTCOMES:
Does early administration of insulin glargine result in a change in hospital length of stay (defined as time between start of insulin infusion and discharge from hospital) when compared to usual care for the treatment of diabetic ketoacidosis? | Until discharge from ICU to general medical unit or from hospital, up to 12 weeks
  Hypothesis: Early administration of insulin glargine will result in shorter hospital length of stay when compared to usual care in patients with DKA.
Does early administration of insulin glargine result in a change in recovery from DKA when compared to usual care for the treatment of diabetic ketoacidosis? | Until discharge from ICU to general medical unit or from hospital, up to 12 weeks
  Recovery defined as blood glucose < 200 and two of: Anion Gap </= 12, Serum Bicarbonate ≥ 15 mEq/L, or pH > 7.3
Does early administration of insulin glargine result in a change in duration of time on IV insulin infusion when compared to usual care for the treatment of diabetic ketoacidosis? | Until discharge from ICU to general medical unit or from hospital, up to 12 weeks
  Hypothesis: Early administration of insulin glargine will result in a shorter duration of time on IV insulin infusion when compared to usual care for the treatment of diabetic ketoacidosis.
Does early administration of insulin glargine result in a change in prevalence of rebound hyperglycemia when compared to usual care for the treatment of diabetic ketoacidosis? | Through 24 hour mark after IV insulin discontinuation
  Rebound hypoglycemia defined as blood glucose > 180 mg/dL in the 24 hours after IV insulin infusion discontinuation
The number of hypoglycemic (defined as blood glucose < 70mg/dL) events occurring while on IV insulin therapy or in the 24h hours after IV insulin infusion discontinuation with early insulin glargine administration compared to usual care | Assessed from time of hospitalization until 24 hour mark after IV insulin discontinuation
  Hypothesis: The occurrence of a hypoglycemic event occurring while on IV insulin therapy or in the 24h hours after IV insulin infusion discontinuation with administration of insulin glargine is comparable to usual care.
The change in mean blood glucose values in the 24 hours and (separately) 48 hours after IV insulin infusion discontinuation | Assessed from time of hospitalization until 48 hour mark after IV insulin discontinuation
  Hypothesis: Early administration of insulin glargine will result in a lower mean value of blood glucose in the 24 and 48 hours after IV insulin infusion discontinuation.
The change in duration of elevated anion gap when compared to usual care | Until discharge from ICU to general medical unit or from hospital, up to 12 weeks
  Hypothesis: Early administration of insulin glargine will result in a shorter duration of elevated anion gap (defined as time with anion gap > 12) when compared to usual care for the treatment of diabetic ketoacidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Adis Keric, PharmD, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with investigators not currently involved in the study.

REFERENCES:
- [Background] Kitabchi AE, Umpierrez GE, Miles JM, Fisher JN. Hyperglycemic crises in adult patients with diabetes. Diabetes Care. 2009 Jul;32(7):1335-43. doi: 10.2337/dc09-9032. No abstract available. PMID 19564476
- [Background] Hirsch IB. Insulin analogues. N Engl J Med. 2005 Jan 13;352(2):174-83. doi: 10.1056/NEJMra040832. No abstract available. PMID 15647580
- [Background] American Diabetes Association. 9. Pharmacologic Approaches to Glycemic Treatment: Standards of Medical Care in Diabetes-2019. Diabetes Care. 2019 Jan;42(Suppl 1):S90-S102. doi: 10.2337/dc19-S009. PMID 30559235
- [Background] Hsia E, Seggelke S, Gibbs J, Hawkins RM, Cohlmia E, Rasouli N, Wang C, Kam I, Draznin B. Subcutaneous administration of glargine to diabetic patients receiving insulin infusion prevents rebound hyperglycemia. J Clin Endocrinol Metab. 2012 Sep;97(9):3132-7. doi: 10.1210/jc.2012-1244. Epub 2012 Jun 8. PMID 22685233
- [Background] Doshi P, Potter AJ, De Los Santos D, Banuelos R, Darger BF, Chathampally Y. Prospective randomized trial of insulin glargine in acute management of diabetic ketoacidosis in the emergency department: a pilot study. Acad Emerg Med. 2015 Jun;22(6):657-62. doi: 10.1111/acem.12673. Epub 2015 May 25. PMID 26013711
- [Background] Houshyar J, Bahrami A, Aliasgarzadeh A. Effectiveness of Insulin Glargine on Recovery of Patients with Diabetic Ketoacidosis: A Randomized Controlled Trial. J Clin Diagn Res. 2015 May;9(5):OC01-5. doi: 10.7860/JCDR/2015/12005.5883. Epub 2015 May 1. PMID 26155506
- [Background] Rappaport SH, Endicott JA, Gilbert MP, Farkas JD, Clouser RD, McMillian WD. A Retrospective Study of Early vs Delayed Home Dose Basal Insulin in the Acute Management of Diabetic Ketoacidosis. J Endocr Soc. 2019 Apr 11;3(5):1079-1086. doi: 10.1210/js.2018-00400. eCollection 2019 May 1. PMID 31069278
- [Background] Gosmanov AR, Gosmanova EO, Dillard-Cannon E. Management of adult diabetic ketoacidosis. Diabetes Metab Syndr Obes. 2014 Jun 30;7:255-64. doi: 10.2147/DMSO.S50516. eCollection 2014. PMID 25061324

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06007508/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT06007508/ICF_001.pdf